CLINICAL TRIAL: NCT04038255
Title: Smartphone Application Versus Group Mindfulness-based Smoking Cessation Intervention for Cancer Patients and Survivors: Reach Versus Effectiveness
Brief Title: Mindfulness Based Smoking Cessation Among Cancer Survivors
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment for the study proved to be a significant challenge, raising important concerns about its overall feasibility.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Taghrid Asfar, Research Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190328
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Smoking
Keywords: cancer; nicotine replacement therapy; mindfulness
MeSH Terms: conditions — Tobacco Smoking; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (Active Comparator): Participants in this group will receive a brief advice to quit smoking, 6-week supplies of nicotine replacement therapy (NRT), and self-help materials to quit smoking.
  Interventions: Drug: Nicoderm C-Q Transdermal Product; Behavioral: Brief advice on quitting smoking; Behavioral: Self-help smoking cessation materials
- Craving-to-Quit app (Experimental): Participants in this group will receive one "in-person" or online orientation session, 6-week supply of NRT, the "Craving-to-Quit" app, and two brief follow-up phone calls.
  Interventions: Drug: Nicoderm C-Q Transdermal Product; Behavioral: Orientation session; Behavioral: Craving-to-Quit app; Behavioral: Two brief follow-up phone calls
- Group Mindfulness Training (Experimental): Participants in this group will receive twice weekly group sessions (eight total during 4 weeks) that were manualized and delivered by instructors experienced in Mindfulness Training (MT) (a single therapist with >4 years of training in MT).
  Interventions: Drug: Nicoderm C-Q Transdermal Product; Behavioral: Orientation session; Behavioral: Group MT sessions

INTERVENTIONS:
Drug: Nicoderm C-Q Transdermal Product — 6 weeks of nicotine replacement therapy patches
Behavioral: Orientation session — This session will occur 2 weeks before quit date. It will be moderated by a certified instructor in MT, and will last approximately 90 min. During the session, participants will learn the purpose, format, and procedures of the study, provide electronic informed consent which will be audio-recorded with their permission, and complete the baseline assessment.
  Arms: Craving-to-Quit app; Group Mindfulness Training
Behavioral: Craving-to-Quit app — The app is comprised of 22 modules for 22 days, 5-15 minutes each, designed to teach MT using audio, video, and animation. The app also includes other features such as social support (quit friend sign-ups, the tip of the week), activity feed (to track interaction with the app), and my morning stats (to track smoking).
  Arms: Craving-to-Quit app
Behavioral: Two brief follow-up phone calls — The first phone call will occur one day before the quit date to remind participants about their quit date and provide support. The second will occur at the end of treatment (around day 60 after quit date) to review progress, provide support, and schedule the 3-month follow-up visit. Each phone call will last approximately 15 minutes.
  Arms: Craving-to-Quit app
Behavioral: Group MT sessions — Total of eight group sessions (twice a week) during 4 weeks. The overarching theme of momentary awareness and acceptance of cravings and affect (e.g., stress, anxiety etc.) will be introduced and reinforced in complementary ways throughout the training. Each session will last 45-60 minutes.
  Arms: Group Mindfulness Training
Behavioral: Brief advice on quitting smoking — Standard advice on how to quit smoking.
  Arms: Usual Care
Behavioral: Self-help smoking cessation materials — Written materials on how to quit smoking including contact info for state tobacco quitline.
  Arms: Usual Care

SUMMARY:
This study will examine the effect of a mindfulness-based smoking cessation program among cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years and older
* Cancer survivors (based on the NCI definition - "a person is considered to be a survivor from the time of diagnosis until the end of life" National Cancer Institute Dictionary of Cancer Terms, 2014)
* Cancer patients currently in active treatment
* Have smoked ≥ 5 cigarettes/day in the past year
* Be interested in making a quit attempt in the next 30 days
* Own a smartphone (apple/android)
* Read/speak English
* Able to consent
* Have no plans to move in the next 3 months
* Are not pregnant or planning to be pregnant in the following 3 months

Exclusion Criteria:

* Have contraindication to NRT (past month myocardial infarction, history of serious arrhythmias/or unstable angina pectoris, dermatological disorder)
* Are currently being treated for a psychiatric condition
* Are currently being treated for smoking cessation, alcoholism, or illicit drug use
* Are adults unable to consent
* Are individuals who are not yet adults
* Are pregnant women
* Are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-28 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taghrid Asfar, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Usual Care Arm was the arm of the intervention where participants would receive a brief advice to quit smoking, 6-week supplies of nicotine replacement therapy, and self-help materials to quit smoking. Unfortunately, the study was closed to enrollment due to difficulty in participant recruitment before we started enrolling to the Usual Care Arm, which would occur after sufficient enrollment in the mindfulness training arm. As a result, no participants were enrolled in the Usual Care Arm.
Period: Overall Study
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Started | 0 | 11 | 9
Completed | 0 | 2 | 3
Not Completed | 0 | 9 | 6
Not completed — Lost to Follow-up | 0 | 9 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study was closed to enrollment due to difficulty in participant recruitment before we started enrolling to the Usual Care Arm; therefore, no participants were enrolled in the Usual Care Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training | Total
Number analyzed (Participants) | 0 | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years, based on the difference between the date of birth provided at baseline compared to the date of consent.
  years |  | 59.40 (15.04) | 64.71 (6.21) | 61.56 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 3 participants that were randomized to a group, but did not complete a baseline; thus we can't verify their gender.
  Participants
    number analyzed (Participants) | 0 | 10 | 7 | 17
    Female |  | 7 | 3 | 10
    Male |  | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 2 | 2 | 4
  Not Hispanic or Latino |  | 8 | 5 | 13
  Unknown or Not Reported |  | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White |  | 6 | 3 | 9
  Non-Hispanic Black |  | 2 | 2 | 4
  Hispanic |  | 2 | 2 | 4
  Asian/Asian American/Pacific Islander |  | 0 | 0 | 0
  Other |  | 0 | 0 | 0
  Unknown/Not Reported |  | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Smoking Abstinence
Description: Number of participants who self-report of not smoking in the past 7-days, not even a puff, confirmed by expired carbon monoxide (CO) level of < 10 ng/ml.
Time Frame: 3 months
Population: Due to difficulties in enrollment, we could not recruit participants for usual care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 11 | 9
Participants
  Self-reported quitting | 0 | 2 | 0
  self-report of quitting confirmed by CO < 10 ng/ml: number analyzed (Participants) | 0 | 2 | 0
  self-report of quitting confirmed by CO < 10 ng/ml | 0 | 1 | 0

2. Secondary Outcome: Change in Number of Cigarettes Smoked Per Day
Description: Self-reported number of cigarettes smoked per day by each participant (Question is: "On average, how many cigarettes do you smoke per day?. Calculated as # of cigarettes reported at Baseline minus # of cigarettes reported at 3-month follow-up)
Time Frame: Baseline, 3 months
Population: Due to difficulties in recruitment, no one was added to Usual Care Arm.
Measure: Mean (Standard Deviation); unit: change in cigarettes/day
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 11 | 9
change in cigarettes/day |  | 0 (0) | 3 (7.55)

3. Secondary Outcome: Number of Participants With Reported Relapse
Description: Relapse is defined as smoking at least once/week on two consecutive weeks.
Time Frame: 3 months
Population: Due to difficulties in recruitment, we were not able to recruit participants for the Usual Care Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 11 | 9
Participants |  | 9 | 9

4. Secondary Outcome: Usability of the Craving-to-Quit App
Description: How usable participants found the app measured by the absolute number of times logged into the app.
Time Frame: 3 months
Population: Only 2 people from the Craving to Quit App arm answered for the 3-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 2 | 0
Participants
  Everyday | 0 | 0 | 0
  Often | 0 | 0 | 0
  Some days | 0 | 2 | 0
  Not often | 0 | 0 | 0
  Not at all | 0 | 0 | 0

5. Secondary Outcome: Usability of the Craving-to-Quit App as Assessed by the Number of Days of Completed App Use
Description: How usable participants found the app measured by self-reported number of completed days for the app.
Time Frame: 3 months
Population: Study was closed to enrollment due to difficulty in participant recruitment before we started enrolling to the Usual Care Arm.We did not have enough people from the Craving-to-Quit arm do the 3-month follow-up to collect or analyze this data.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 2 | 0
Participants
  Every day |  | 0 |
  Often |  | 0 |
  Some days |  | 2 |
  Not often |  | 0 |
  Not at all |  | 0 |

6. Secondary Outcome: Usability of the Craving-to-Quit App as Assessed by the Comfortability With the App
Description: How usable participants found the app measured by the comfortability of the app via questionnaire with scores ranging from 0-10 with the higher score indicating increased comfortability with the app.
Time Frame: 3 months
Population: Number of participants from this treatment arm who responded to the 3-month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mindfulness Training: Participants in this group will receive twice weekly group sessions (eight total during 4 weeks) that were manualized and delivered by instructors experienced in Mindfulness Training (MT) (a single therapist with >4 years of training in MT).
  Nicoderm C-Q Transdermal Product: 6 weeks of nicotine replacement therapy patches
  Orientation session: This session will occur 2 weeks before quit date. It will be moderated by a certified instructor in MT, and will last approximately 90 min. During the session, participants will learn the purpose, format, and procedures of the study, provide electronic informed consent which will be audio-recorded with their permission, and complete the baseline assessment.
  Group MT sessions: Total of eight group sessions (twice a week) during 4 weeks. The overarching theme of momentary awareness and acceptance of cravings and affect (e.g., stress, anxiety etc.) will be introduced and reinforced in complementary ways throughout the training. Each session will last 45-60 minutes.
Arm/Group | Usual Care | Craving-to-Quit App | Mindfulness Training
Number analyzed (Participants) | 0 | 2 | 0
units on a scale |  | 10 (0) |

7. Secondary Outcome: Acceptability
Description: Assessed by 3 items "How satisfied were you with the intervention?", "How likely are you to recommend this intervention to a friend?" and "How useful was the intervention?" Each question is scored from 0-10 with the higher score indicating increased acceptability.
Time Frame: 3 months
Population: Study was closed to enrollment due to difficulty in participant recruitment before we started enrolling to the Usual Care Arm. Only 5 people answered the 3 month follow-up for their corresponding groups (2 for Craving to Quit, 3 for Group Mindfulness Training).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 2 | 3
score on a scale
  How satisfied were you with the intervention? |  | 7.5 (0.71) | 9 (1.73)
  How likely are you to recommend this intervention to a friend? |  | 10 (0) | 10 (0)
  How useful was the intervention |  | 10 (1.41) | 10 (0)

8. Secondary Outcome: Feasibility of Recruitment as Assessed Via Enrollment Rate
Description: Percentage of enrolled in each arm out of the 44 that were originally recruited (number recruited divided by number enrolled multiplied by 100). A feasible recruitment is defined as an enrollment rate of 70% or higher.
Time Frame: Baseline
Population: Study was closed to enrollment due to difficulty in participant recruitment before we started enrolling to the Usual Care Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 44 | 44
Participants |  | 11 | 9

9. Secondary Outcome: Attrition
Description: Defined as the number of participants not having a final visit at the end of treatment, categories include mortality, withdrawal from the study, transfer to non-study clinics, loss to follow-up without identifiable cause.
Time Frame: 3 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
Number analyzed (Participants) | 0 | 11 | 9
participants
  Loss to follow-up without identifiable cause |  | 9 | 5
  Mortality |  | 0 | 0
  Withdrawal |  | 0 | 1
  Transfer to non-study clinic |  | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Study was closed to enrollment due to difficulty in participant recruitment before we started enrolling to the Usual Care Arm. There were no participants assigned to the Usual Care Arm; therefore, the at-risk number is zero for this arm.
Arm/Group | Usual Care | Craving-to-Quit App | Group Mindfulness Training
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/0 | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT04038255/Prot_SAP_000.pdf